CLINICAL TRIAL: NCT03715140
Title: Evaluation of the Crucumin Effects on the Cellular and Humoral Immune Systems in Osteoarthritis Patients; a Randomised Double Blind Placebo Control Clinical Trial
Brief Title: Crucumin Effects on the Immune System in Osteoarthritis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Mojgan Mohammadi, Associate Professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.MUMS.MEDICAL.REC.1397.118
Record Dates: First submitted 2018-10-15; First posted 2018-10-23 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Crucumin, Flowcytometry
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who will recieve crucumin (Experimental): patients who prescribing crucumin 80 mg daily for three months will be evaluated. A sample will be taken before taking the drug.
  Interventions: Drug: Crucumin
- Patients who will receive placebo (Placebo Comparator): Patients who prescribing placebo daily for three months will be evaluated. A sample will be taken before taking the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Crucumin — Evaluation of the effect of Crucumin in patients with osteoarthritis
  Other Names: nanocrucumin
  Arms: Patients who will recieve crucumin
Drug: Placebo — Placebo
  Other Names: Crucumin placebo
  Arms: Patients who will receive placebo

SUMMARY:
In this study, the effects of crucumin on cellular and humoral immune system in patients with osteoarthritis will be investigated. Concentration of CXCL8, April, CX3CL1 and IL-17 will be evaluated with ELISA. TH-1, TH-17, TReg and Ly.B cells count will be measured by Flowcytometry. MicroRNA-720, MicroRNA-155, MicroRNA-16 and MicroRNA-146a gene expression will be measured with Real Time PCR technique.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effect of the active ingredient of crucumin on the reduction of symptoms of osteoarthritis. Of the 30 patients participating in this study, a blood sample will be taken at the beginning of the study, and then after three months of taking the crucumin. To evaluate the response to treatment, after each person sampling, we will analyze cell count for Th-1, Th-17, TReg and Ly.B by flowcytomtry method. Also we will measure cytokines level of IL-17, CXCL8, CX3CL1 and April by ELISA method. Finally we evaluate the gene expression of MicroRNA-720, MicroRNA-155, MicroRNA-146a and MicroRNA-16 by Real Time PCR technique.

ELIGIBILITY:
Inclusion Criteria:

Osteoarthritis patients who have been diagnosed with a rheumatologist physician based on clinical examinations and laboratory tests

Exclusion Criteria:

Affected by any other acute or chronic underlying disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09-21 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
IL-17 | Baseline
  Cytokine level

SECONDARY OUTCOMES:
IL-17 | Baseline and three months
  Cytokine level
TH-1 | Baseline and three months
  Cell counting
MicroRNA-720 | Baseline and three months
  Gene expression
CXCL8 | Baseline and three months
  Cytokine level
CXCL1 | Baseline and three months
  Cytokine level
April | Baseline and three months
  Cytokine level
TH-17 | Baseline and three months
  Cell counting
TReg | Baseline and three months
  Cell counting
Ly.B | Baseline and three months
  Cell counting
MicroRNA-155 | Baseline and three months
  Gene expression
MicroRNA-146a | Baseline and three months
  Gene expression
MicroRNA-16 | Baseline and three months
  Gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Mojgan Mohammadi, Ph.D, Principal Investigator — Department of Immunology, Faculty of Medicine, Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Mahdi Atabaki, Mashhad, Iran

IPD SHARING:
Plan to Share IPD: Undecided
Preferring the data to remain confidential